CLINICAL TRIAL: NCT05066451
Title: Demonstration and Comparison of 5% Dextrose Prolotherapy and 15% Dextrose Prolotherapy Efficacy in Lateral Epicondylitis
Brief Title: 5% and 15% Dextrose Prolotherapy Efficacy in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FTRTEZTASKIN
Record Dates: First submitted 2021-09-20; First posted 2021-10-04 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; dextrose prolotherapy; pain; injection
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- %5 dextrose prolotherapy (Experimental): A total of 3 sessions of prolotherapy solution containing 5% dextrose will be applied at the beginning, 3rd week, and the 6th week.
  Interventions: Other: %5 dextrose prolotherapy
- %15 dextrose prolotherapy (Active Comparator): A total of 3 sessions of prolotherapy solution containing 15% dextrose will be applied at the beginning, 3rd week, and the 6th week.
  Interventions: Other: %15 dextrose prolotherapy

INTERVENTIONS:
Other: %5 dextrose prolotherapy — Patients in the study group will receive a total of 3 sessions of prolotherapy solution containing 5% dextrose at the beginning(0.) 3rd week and 6th week.
  Prolotherapy was planned with the multiplanar injection technique (peppering technique) after palpating the most sensitive point on the lateral epicondyle and entering the lateral epicondyle from here and ensuring bone contact.
  Arms: %5 dextrose prolotherapy
Other: %15 dextrose prolotherapy — Patients in the study group will receive a total of 3 sessions of prolotherapy solution containing 15% dextrose at the beginning(0.) 3rd week and 6th week.
  Prolotherapy was planned with the multiplanar injection technique (peppering technique) after palpating the most sensitive point on the lateral epicondyle and entering the lateral epicondyle from here and ensuring bone contact.
  Arms: %15 dextrose prolotherapy

SUMMARY:
In the treatment of lateral epicondylitis, 5% dextrose prolotherapy is aimed to be more reliable than 15% prolotherapy in terms of side effects and to show that it is similar in terms of efficacy in treatment.

DETAILED DESCRIPTION:
For this prospective randomized controlled study, volunteer patients who met the inclusion criteria and applied to the Health Sciences University, Istanbul Physical Therapy and Rehabilitation Training and Research Hospital, Physical Medicine and Rehabilitation Outpatient Clinic will be included in the study. Participants who volunteered for the study will be divided into study groups and control groups by stratified randomization. A total of 26 volunteers will be recruited.

A solution to be used for prolotherapy is containing 30% dextrose, 2% lidocaine, and physiological saline.

In the beginning, all patients were asked about gender, age, body mass index, education level, occupation, duration of complaint, dominant side and affected extremity, previous treatments, and when the last treatment was applied.

Patients in the study group will receive a total of 3 sessions of prolotherapy solution containing 5% dextrose at the beginning(0.) 3rd week and 6th week.

Prolotherapy was planned with the multiplanar injection technique (peppering technique) after palpating the most sensitive point on the lateral epicondyle and entering the lateral epicondyle from here and ensuring bone contact.

Patients in the control group will receive a total of 3 sessions of prolotherapy solution containing 15% dextrose, initially (0.) Week 3 and Week 6. The injection will be made with the same method as the study group.

Measurements; will be evaluated at baseline (week 0), immediately after treatment at Week 3, Week 6, and Week 12.

Patients; In the evaluation of the visual analog scale (VAS), quick Disabilities of the Arm, Shoulder and Hand (QDASH), Grip strength, hand dynamometer measurements, and adverse events during the study period will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Pain score ≥3 according to VAS for more than 3 months in the lateral elbow joint
* tenderness on palpation over the lateral epicondyle
* Positiveness in at least two of the tests specific to lateral epicondylitis(LE) (Mills test, resistant middle finger extension and cozen test),
* > 20 years old , < 60 years old

Exclusion Criteria:

* Patients who received physical therapy modalities and/or steroid injections in the last 3 months,
* Having a history of malignancy,
* Pregnant cases,
* Those who have bone and joint diseases in the neck, shoulder and elbow,
* Patients with infection in the treatment area,
* Patients with arrhythmia or pacemaker in the heart,
* Patients receiving coagulation disorder or anticoagulant therapy,
* Those with local dermatological problems,
* Patients with a history of surgery in the elbow joint,
* Having a tendon tear
* Presence of nerve involvement
* Lack of cooperation and refusal to participate in the study due to cognitive dysfunction

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
The upper extremity disability level | Change from baseline upper extremity disability level at 3, 6, and 12 weeks
  The upper extremity disability level will be evaluated by using the Quick Disabilities of Arm, Shoulder and Hand (QDASH) scale. The maximum score is 100 points. A higher score indicates a worse disability level.
Pain intensity | Change from baseline pain intensity at 3, 6, and 12 weeks
  Pain intensity will be evaluated by using a visual analog scale (VAS). The maximum score is 10 points. A higher score indicates a worse pain level.

SECONDARY OUTCOMES:
Hand grip strength | Change from baseline hand grip strength at 3, 6, and 12 weeks
  The standard evaluation tool (a hand dynamometer) will used for measuring grip and squeeze strength minimum value 0 and there is not maximum value, bigger values mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Taskin, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospita; Fatma Nur Kesiktas, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospita
Locations (1):
- İstanbul physical medicine rehabilitation training &research hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fornalski S, Gupta R, Lee TQ. Anatomy and biomechanics of the elbow joint. Tech Hand Up Extrem Surg. 2003 Dec;7(4):168-78. doi: 10.1097/00130911-200312000-00008. PMID 16518218
- [Background] Kahlenberg CA, Knesek M, Terry MA. New Developments in the Use of Biologics and Other Modalities in the Management of Lateral Epicondylitis. Biomed Res Int. 2015;2015:439309. doi: 10.1155/2015/439309. Epub 2015 May 31. PMID 26114106
- [Background] Rabago D, Slattengren A, Zgierska A. Prolotherapy in primary care practice. Prim Care. 2010 Mar;37(1):65-80. doi: 10.1016/j.pop.2009.09.013. PMID 20188998
- [Background] Jensen KT, Rabago DP, Best TM, Patterson JJ, Vanderby R Jr. Early inflammatory response of knee ligaments to prolotherapy in a rat model. J Orthop Res. 2008 Jun;26(6):816-23. doi: 10.1002/jor.20600. PMID 18240327